CLINICAL TRIAL: NCT04384224
Title: The Clinical Benefits of the Combination Use of Acupuncture and Antihistamine on Trigeminal Neuralgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH109-REC3-007
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- sham acupuncture + placebo tablet group (Placebo Comparator): sham acupuncture point + placebo tablet
  Interventions: Other: acupuncture
- true acupuncture + placebo tablet group (Experimental): true acupuncture point + placebo tablet
  Interventions: Other: acupuncture
- true acupuncture + antihistamine group (Experimental): true acupuncture point + Dexchlorpheniramine (4 mg)
  Interventions: Other: acupuncture
- sham acupuncture + antihistamine group (Sham Comparator): sham acupuncture point + Dexchlorpheniramine (4 mg)
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — use disposable sterile steel needles to insert to the acupuncture point

SUMMARY:
Trigeminal neuralgia is a paroxysmal extreme pain and is an unmet clinical need, we hope that our discovery about the antihistamine and acupuncture can be used in the treatment trigeminal neuralgia. This present study aims to further investigate whether antihistamine dexchlorpheniramine can facilitate the analgesic effect of acupuncture in patients with trigeminal neuralgia.

DETAILED DESCRIPTION:
Trigeminal neuralgia is a paroxysmal extreme pain that occurs in the region dominated by facial trigeminal nerve. It is characterized by repetition and irregularity. Once the disease occurs, the pain is generally unbearable. Carbamazepine or other drugs is the main treatment methods. However, most patients will experience side effects so that drug treatments for trigeminal neuralgia has its limitation limitation. Surgical treatments have better efficacy but with greater risk.

The efficacy of acupuncture for pain treatment has been widely demonstrated by many clinical trials. A recent meta analysis has demonstrated that significant differences of efficacy between true and sham acupuncture indicate that acupuncture is more than a placebo. However, there are few clinical randomized controlled trials reporting the efficacy of acupuncture on trigeminal neuralgia.

Histamine H1 receptor antagonists are commonly used for treating allergy. Recently, we found that histamine H1 receptor antagonists at relatively low doses facilitate electroacupuncture (EA) analgesia in the acetic acid-induced abdominal writhing test. We have also conducted a clinical trial to demonstrate that H1 receptor antagonists facilitate EA analgesia in healthy volunteers. The study recruited 40 healthy normal subjects we found that EA at bilateral ST36 and GB34 plus high-dose dexchlorpheniramine (4 mg) produced greater pain threshold increases as than EA alone groups, suggesting the combination use of H1 antihistamine can facilitate acupuncture analgesia in humans.

This study aims to investigate whether antihistamine dexchlorpheniramine can also facilitate the analgesic effect of acupuncture in patients with trigeminal neuralgia. The experimental design is as follows: This experiment will recruit 40 healthy subjects, randomly divided into 4 groups, each group of 10 patients (1) sham acupuncture + placebo tablet group, (2) true acupuncture + placebo tablet group , (3) true acupuncture + antihistamine group and (4) sham acupuncture + antihistamine group. The treatment duration is one week for 3 acupuncture/sham acupuncture treatment. Dexchlorpheniramine (4 mg) or placebo tablets will be administered at the sleeping time the day before acupuncture treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 20 2. Occurrence of episodes of intense facial paroxysmal pain in territory innervated by the trigeminal nerve (VAS score ≥ 6) 3. Presence of a normal neurologic examination 4. Neurologist confirm- Normal neuroimaging analysis 5. Duration of each pain episode < 15 minutes

Exclusion Criteria:

* 1. Patient refuse to participate 2. Psychologic instability 3. Atypical pain location (eg, no specific trigger points) 4. Anticlotting therapy 5. Secondary trigeminal neuralgia

  * Multiple sclerosis
  * Temporomandibular joint disorders
  * Neoplasias 6. Altered neurologic profile
  * Hypoesthesia
  * Dysesthesia
  * Anesthesia
  * Paresis 7. Association with other cranial nerve neuralgias (eg, glossopharyngeal neuralgia) 8. Imagiologic alterations 9. Proposed surgical intervention
  * Compression of the Gasser ganglion
  * Micro vascular decompression
  * Radiofrequency rhizotomy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
The change of Visual Analogue Scale | evaluated at the beginning of the treatment (day 0), the treatment day (3 session per week; just after treatment), and Day 21 (3 weeks) after the end of the treatment (follow-up)
  Patients located their relative pain in a line marked in each extremity with 0 (0: no pain-on the left) and 10 (10: the worst pain imaginable-on the right)

SECONDARY OUTCOMES:
Short Form Health Survey-36 | evaluated at the beginning of the treatment (day 0) and Day 21 (3 weeks) after the end of the treatment (follow-up)
  a 36-item questionnaire assessing functional health and well-being during the previous month. Testing of the Taiwanese version has demonstrated validity similar to that of other language versions. The SF-36 evaluates quality of life in 8 domains: physical functioning (PF), role limitations due to physical problems (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role limitations due to emotional problems (RE), and general mental health (MH). Five of the scales (PF, RP, BP, SF and RE) indicate the absence of limitations or disability. The remaining 3 scales (GH, VT and MH) indicate a positive state of well-being, with mid-range scores indicating no reported limitations or disabilities. In this study, items in each domain will be aggregated and transformed into a scale from 0 to 100, with higher scores indicating better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chen Lee, Study Director — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No